CLINICAL TRIAL: NCT07230860
Title: A Phase 2b, Multicenter, Randomized, Double-blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Efficacy and Safety of JNJ-95597528 for the Treatment of Adult Participants With Moderate to Severe Atopic Dermatitis
Brief Title: A Study of JNJ-95597528 in Participants With Moderate to Severe Atopic Dermatitis
Acronym: READY-AD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 95597528ADM2001; 95597528ADM2001 (Other: Janssen Research & Development, LLC); 2025-523464-20-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1: JNJ-95597528 (Dose 1) (Experimental): Participants will receive JNJ-95597528 Dose 1 on Weeks 0, 2, 12, and 24.
  Interventions: Drug: JNJ-95597528
- Group 2: JNJ-95597528 (Dose 2 and 3) (Experimental): Participants will receive JNJ-95597528 Dose 2 on Week 0 followed by JNJ-95597528 Dose 3 on Weeks 12, and 24.
  Interventions: Drug: JNJ-95597528
- Group 3: JNJ-95597528 (Dose 4 and 5) (Experimental): Participants will receive JNJ-95597528 Dose 4 on Week 0 followed by JNJ-95597528 Dose 5 on Weeks 12, and 24.
  Interventions: Drug: JNJ-95597528
- Group 4: Placebo and JNJ-95597528 (Dose 2 and 3) (Placebo Comparator): Participants will receive placebo from Weeks 0 to 12 , then switch to receive JNJ-95597528 Dose 2 administered at Week 12 followed by Dose 3 at Week 24.
  Interventions: Drug: JNJ-95597528; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-95597528 — JNJ-95597528 will be administered subcutaneously.
Drug: Placebo — Placebo will be administered subcutaneously.
  Arms: Group 4: Placebo and JNJ-95597528 (Dose 2 and 3)

SUMMARY:
The purpose of this study is to assess how well JNJ-95597528 works compared to placebo in participants with moderate to severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion criteria:

* Be otherwise healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening
* Meets all the following disease activity criteria: a. Chronic atopic dermatitis (AD), according to American Academy of Dermatology Consensus Criteria with onset of symptoms at least 1 year prior to screening visit; b. Eczema area and severity index (EASI) score greater than or equal to (>=) 16 at the screening and Week 0; c. validated investigator global assessment for atopic dermatitis (vIGA-AD) score >= 3 at screening and Week 0; d. >= 10% body surface area (BSA) of AD involvement at screening and Week 0; e. Documented history (within 6 months before screening) of either inadequate response or inadvisability to medicated topical treatments for AD or inadequate response to systemic therapies (within 12 months before screening)
* Must sign an informed consent form (ICF) indicating that the participant understands the purpose of, and procedures required for, the study and is willing to participate in the study
* If willing to participate in the substudy, must sign a separate ICF for the corresponding substudy (or substudies)
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, lifestyle restrictions, and other study procedures

Exclusion criteria:

* History of substance abuse or alcohol abuse within 1 year before screening
* In the investigator's opinion, any clinically significant results from the 12-lead ECG, chemistry, hematology, or urinalysis laboratory tests obtained at the screening visit that would affect interpretation of study data or the participant's safety in the study
* Known or suspected immunodeficiency, including history of invasive opportunistic infections
* Previously received JNJ-95597528
* Has known hypersensitivity or intolerance to JNJ-95597528 or its excipients or to any biologic medication or known allergies, or clinically significant reactions to murine, chimeric, monoclonal antibodies (mAbs), or antibody fragments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-02-13 (Estimated); Primary Completion 2026-11-19 (Estimated); Study Completion 2028-02-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with Eczema Area and Severity Index (EASI) 75 Response at Week 12 | Week 12
  EASI-75 response is defined as at least 75 percent (%) improvement from baseline in EASI total score. EASI is a validated measure used to assess the severity and extent of AD with scores ranging from 0 to 72. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) will each be assessed for severity by the investigator or designee on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement will be assessed as a percentage by body area of head, trunk, upper limbs, and lower limbs, and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). Here higher score indicates higher severity of AD.

SECONDARY OUTCOMES:
Proportion of Participants with EASI 90 Response at Week 12 | Week 12
  EASI-90 response is defined as at least 90% improvement from baseline in EASI total score. EASI is a validated measure used to assess the severity and extent of AD with scores ranging from 0 to 72. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) will each be assessed for severity by the investigator or designee on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement will be assessed as a percentage by body area of head, trunk, upper limbs, and lower limbs, and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). Here higher score indicates higher severity of AD.
Proportion of Participants with EASI 100 Response at Week 12 | Week 12
  EASI-100 response is defined as at least 100% improvement from baseline in EASI total score. EASI is a validated measure used to assess the severity and extent of AD with scores ranging from 0 to 72. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) will each be assessed for severity by the investigator or designee on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement will be assessed as a percentage by body area of head, trunk, upper limbs, and lower limbs, and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). Here higher score indicates higher severity of AD.
Percent Change from Baseline in EASI Total Score at Week 12 | Baseline, Week 12
  Percent change from baseline in EASI total score will be reported. EASI is a validated measure used to assess the severity and extent of AD with scores ranging from 0 to 72. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) will each be assessed for severity by the investigator or designee on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement will be assessed as a percentage by body area of head, trunk, upper limbs, and lower limbs, and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). Here higher score indicates higher severity of AD.
Proportion of Participants with Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) Score of 0 or 1 and a Reduction of >= 2 Points from Baseline, at Week 12 | Week 12
  Proportion of participants with vIGA-AD score of 0 or 1 and a reduction of >=2 points from baseline at Week 12 will be reported. vIGA-AD is an assessment instrument used in clinical studies to rate the severity of AD, based on a 5-point scale ranging from 0 (clear) to 4 (severe). The IGA score is selected using the morphological descriptors that best describe the overall appearance of the AD lesions at a given time point. Higher scores are indicative of a more severe AD.
Proportion of Participants with vIGA-AD Score of 0 and a Reduction of >= 2 points from Baseline, at Week 12 | Week 12
  Proportion of participants with vIGA-AD score of 0 and a reduction of >=2 points from baseline at Week 12 will be reported. vIGA-AD is an assessment instrument used in clinical studies to rate the severity of AD, based on a 5-point scale ranging from 0 (clear) to 4 (severe). The IGA score is selected using the morphological descriptors that best describe the overall appearance of the AD lesions at a given time point. Higher scores are indicative of a more severe AD.
Proportion of Participants with >= 4-Point Improvement in Peak Pruritus Numeric(al) Rating Scale (PP-NRS) from Baseline, at Week 12 | Week 12
  Proportion of participants with >=4-point improvement from baseline in PP-NRS scale at Week 12 will be reported. PP-NRS is a single item asking participants to assess their worst itch over the past 24 hours. There are 11 response categories, ranging from 0 (no itch) to 10 (worst itch imaginable). Higher score indicates greater severity.
Percent Change from Baseline in PP-NRS Score at Week 12 | Baseline, Week 12
  Percent change from baseline in PP-NRS score will be reported. PP-NRS is a single item asking participants to assess their worst itch over the past 24 hours. There are 11 response categories, ranging from 0 (no itch) to 10 (worst itch imaginable). Higher score indicates greater severity.
Percent Change from Baseline in Score of Item 2 of Atopic Dermatitis Sleep Scale (AD Sleep Scale) at Week 12 | Baseline, Week 12
  Percent change from baseline in the score of Item 2 of AD Sleep Scale at Week 12 will be reported. The AD Sleep Scale is a validated 3-item participant-reported outcome (PRO) instrument to capture self-reported impact of itch on sleep disturbance each day, including difficulty falling asleep, number of night-time awakenings, and difficulty falling back asleep after waking during the previous night. For Item 2, participants select the number of times they woke up each night, ranging from 0 to 29 times. Higher score indicates more sleep disturbance.
Proportion of Participants with >= 4 Point Improvement in Skin Pain Numeric Rating Scale (Skin Pain NRS) from Baseline, at Week 12 | Week 12
  Proportion of participants with >= 4 point improvement from baseline in skin pain NRS at Week 12 will be reported. Skin Pain NRS is a single item asking participants to assess their worst skin pain over the past 24 hours. There are 11 response categories, ranging from 0 (no pain) to 10 (worst pain imaginable). Higher score indicates more pain.
Percent Change from Baseline in Skin Pain NRS at Week 12 | Baseline, Week 12
  Percent change from baseline in Skin Pain NRS at Week 12 will be reported. Skin Pain NRS is a single item asking participants to assess their worst skin pain over the past 24 hours. There are 11 response categories, ranging from 0 (no pain) to 10 (worst pain imaginable). Higher score indicates more pain.
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to approximately Week 12
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the intervention. TEAEs are AEs with onset during the intervention phase or that are a consequence of a preexisting condition that has worsened since baseline. An SAE is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product and is medically important.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency